CLINICAL TRIAL: NCT03087903
Title: A Phase 2 Study of Grape Seed Extract (GSE) Product in Asymptomatic Non-Metastatic Prostate Cancer Patients With Rising Prostate Specific Antigen (PSA)
Brief Title: A Study of Grape Seed Extract in Asymptomatic Non-Metastatic Prostate Cancer Patients With Rising PSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Cancer League of Colorado (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-0607.cc
Record Dates: First submitted 2017-03-13; First posted 2017-03-23 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
Keywords: Prostate Specific Antigen (PSA); Non-Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Grape Seed Extract; leucoselect phytosome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 150 mg of Grape Seed Extract (GSE) (Experimental): 150 mg of GSE twice daily in the form of 75 mg capsule of Leucoselect Phytosome preparation.
  Interventions: Dietary Supplement: Grape Seed Extract

INTERVENTIONS:
Dietary Supplement: Grape Seed Extract — Patients will take 150 mg of Grape Seed Extract (GSE) product by mouth twice daily (in the form of 75 mg capsule of Leucoselect Phytosome preparation). Total oral dosage is 300 mg of GSE per day for one year. Patients will be evaluated every 6 weeks for 3 months, then every 3 months thereafter for up to one year. PSA measurements will be obtained at these scheduled visits.
  Other Names: Leucoselect Phytosome

SUMMARY:
Patients will take 150 mg of GSE product by mouth twice daily and will be evaluated every 6 weeks for 3 months, then every 3 months thereafter for up to one year.

DETAILED DESCRIPTION:
Patients will take 150 mg of GSE product by mouth twice daily in the form of 75 mg capsule of Leucoselect Phytosome preparation; total oral dosage is 300 mg GSE per day for one year. Patients will be evaluated every 6 weeks for 3 months, then every 3 months thereafter for up to one year. PSA measurements will be obtained at these scheduled visits and patients must not have a doubling of their PSA (compared to baseline) by 3 months in order to continue on study. Patients who meet criteria to continue on study will be treated until disease progression or for one year (whichever comes first).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent has been obtained.
2. Adults > or = 18 years of age.
3. Histologically confirmed prostate adenocarcinoma.
4. Evidence of rising PSA, on 2 separate occasions, at least one week apart. Baseline PSA must be ≥ 0.2 ng/mL at the time of screening. Radiographic evidence of disease is not allowed.
5. Patients must have sufficient PSA time points prior to enrollment (a minimum of 3 PSA levels within a six month period) to calculate a baseline PSA doubling time.
6. Patients must not be on active LHRH agonist/antagonist therapy and must have testosterone level > 50 ng/dL.
7. Patients must not be on active anti-androgen therapy or 5-alpha reductase inhibitors. Patients on stable dose of 5-alpha reductase inhibitors for benign prostatic hypertrophy for at least 12 months may continue. They must withdraw from the study if this is stopped while on study.
8. Patients who are candidates for local salvage therapy must have had this option pursued or discussed; and the patient must have either declined salvage therapy or was deemed not to be a candidate for salvage therapy.
9. Patients who have PSA recurrence after local salvage therapy may participate in this study.
10. Patients with hormone sensitive disease who received prior androgen deprivation therapy as part of primary/salvage local treatment or patients receiving intermittent androgen deprivation therapy will be allowed to participate.
11. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
12. Adequate hematologic function (absolute neutrophil count [ANC]≥1,500 cells/µL; hemoglobin ≥9 g/dL, platelets ≥75,000/µL).
13. Adequate renal function (serum creatinine ≤ 2X the upper limit of normal (ULN)
14. Adequate hepatic function (total bilirubin ≤ 2 x upper limit of normal [ULN], alanine aminotransferase [ALT]≤ 3xULN, aspartate aminotransferase [AST]≤3 x ULN).
15. Patients can continue taking what they are taking at the time they start on the study, but agree not to start any new (over the counter) herbal supplement on regular basis during study duration.
16. Prior chemotherapy for prostate cancer (upfront, adjuvant, etc.) is allowed as long as it was not given for hormone-refractory disease.

Exclusion Criteria:

1. Patients who are on active surveillance for untreated localized disease may not participate in this study.
2. Inability to swallow gelatin capsules, or any medical condition that interferes with normal gastrointestinal absorption.
3. Major surgery, radiation, or treatment with any other investigational drug within 2 weeks of study treatment.
4. Documented hypersensitivity reaction to any product with GSE (see complete list in Appendix 1).
5. Known chronic infection with human immunodeficiency virus (HIV) or viral hepatitis.
6. Symptomatic prostate cancer as determined by cancer-related pain requiring narcotic pain medication.
7. History of another cancer is exclusionary unless it is believed to be likely cured or is unlikely to be fatal in the next 3 years (e.g. squamous cell carcinoma, superficial bladder cancer, chronic lymphocytic leukemia, etc).
8. Very fast PSA doubling time of less than 4 weeks, if the absolute PSA is > 2 ng/mL.
9. Known allergy/intolerance to soy, phosphatidycholine or any other constituents of grape seed extract.

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
The number of patients with PSA response | 6 weeks and 3, 6, 9, and 12 months
  PSA response will be defined as an increase in prostate specific antigen (PSA) doubling time (PSADT) of 30% (PSADT is the length of time it takes for a PSA to double based on an exponential growth pattern). Patients must have a PSA level of ≥ 0.2 at study entry and should have at least three prior PSA values with dates from which to calculate a PSA doubling time.

SECONDARY OUTCOMES:
The rate of change of the PSA over time (PSA velocity) for each patient | 6 weeks and 3, 6, 9, and 12 months
  PSA velocity will be calculated as a change from the first PSA reading, standardized as PSA change per month. PSA Response will be defined as increase in PSADT of 30% (PSADT is the length of time it takes for a PSA to double based on an exponential growth pattern). Biomarkers will be defined as proinflammatory cytokines, lipid and comprehensive metabolic panel in patient serum samples as well as, gut microbiome (measured by by high-throughput16S sequencing), plasma and stool metabolomics (after short and long-term consumption of GSE), and the effects of diet on gut microbiome.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Maroni, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Cancer Center, Aurora, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado

IPD SHARING:
Plan to Share IPD: No